CLINICAL TRIAL: NCT04153760
Title: A Pilot Study Assessing the Feasibility of a Randomized Controlled Trial Evaluating Aspirin in Postpartum Women at Risk of Developing Venous Thromboembolism
Brief Title: Pilot PARTUM Trial: Postpartum Aspirin to Reduce Thromboembolism Undue Morbidity
Acronym: PARTUM
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Venous Thromboembolism Clinical Trials and Outcomes Research (CanVECTOR) Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: REB19-1237
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Venous Thromboembolism; Postpartum Period; Aspirin
Keywords: deep vein thrombosis; pulmonary embolism; postpartum; pregnancy; thrombophilia; cesarean delivery; pre-eclampsia; postpartum hemorrhage
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism; Thrombophilia; Pre-Eclampsia; Postpartum Hemorrhage | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin (Active Comparator): Aspirin 81 mg daily for six weeks post-randomization (postpartum)
  Interventions: Drug: Aspirin 81 mg
- Placebo (Placebo Comparator): Placebo daily for six weeks post-randomization (postpartum)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin 81 mg — Aspirin 81 mg p.o. daily
  Other Names: acetylsalicylic acid; ASA
  Arms: Aspirin
Drug: Placebo — Placebo p.o. daily
  Arms: Placebo

SUMMARY:
The pilot PARTUM trial is a randomized, multicenter, placebo-controlled trial. Women who are at modest risk of VTE (as defined by the inclusion criteria) will be identified during pregnancy, labor and delivery and up to 48 hours postpartum. Eligible and consenting participants will be randomly assigned to one of two study arms: aspirin 81 mg daily or placebo daily for 6 weeks.

DETAILED DESCRIPTION:
The purpose of the pilot PARTUM trial is to determine whether it is feasible to conduct a larger randomized controlled trial to determine whether low-dose aspirin is efficacious and safe at preventing postpartum venous thromboembolism (VTE) in women at increased risk of VTE, compared to placebo.

Given the large sample size needed to adequately power a large multicenter trial that assesses the efficacy of aspirin 81 mg versus placebo, the investigators first need to determine if it is possible to recruit enough women. If the pilot trial is successful and there are no major changes to the study design, then the secondary clinical outcomes collected in the pilot trial will be used in the analysis of the full multicenter trial.

ELIGIBILITY:
Inclusion Criteria: Study inclusion criteria includes one (or more) first order criterion or two (or more) second order criteria. A patient is still eligible if they have multiple criteria met, at the discretion of the local investigator.

ONE (or more) First Order Criteria:

1. Known inherited thrombophilia diagnosed prior to enrolment:

   i) Heterozygous factor V Leiden, OR ii) Heterozygous prothrombin gene variant, OR iii) Protein C deficiency, OR iv) Protein S deficiency
2. Immobilization (90% of waking hours spent in bed) for ≥7 days anytime during the antepartum period

TWO (or more) Second Order Criteria:

1. Postpartum infection
2. Postpartum hemorrhage (>1000 mL of blood loss, regardless of delivery mode)
3. Pre-pregnancy BMI ≥30 kg/m2
4. Emergency or unplanned cesarean delivery
5. Smoking ≥5 cigarettes/day before pregnancy
6. Pre-eclampsia
7. Current pregnancy ending in stillbirth (pregnancy loss >20 weeks gestation)
8. Small-for-gestational-age infant (<3rd percentile adjusted for gestational age and sex).
9. Previous history of superficial vein thrombosis

Exclusion Criteria:

1. More than 48 hours since delivery
2. Received more than 2 doses of low-molecular-weight heparin (LMWH) since delivery
3. Need for postpartum LMWH prophylaxis or systemic anticoagulation as judged by the local investigator. May include but is not limited to:

   1. Documented history of provoked or unprovoked VTE
   2. Mechanical heart valve(s)
   3. Known antiphospholipid syndrome
   4. Known high-risk inherited thrombophilia i) Antithrombin deficiency; ii) Homozygous factor V Leiden; iii) Homozygous prothrombin gene mutation; iv) Compound heterozygosity factor V Leiden and prothrombin gene mutation; v) More than one inherited thrombophilia
4. Need for postpartum aspirin as judged by the local investigator. May include but is not limited to:

   1. Documented history of myocardial infarction
   2. Documented history of ischemic stroke or transient ischemic attack (TIA)
5. Contraindication to aspirin including:

   1. History of known aspirin allergy
   2. Documented history of a gastrointestinal ulcer
   3. Known platelet count <50 x 109/L at any time during the current pregnancy or postpartum
   4. Active bleeding at any site, excluding normal vaginal bleeding, at the time of randomization
   5. Most recent known hemoglobin ≤70 g/L documented during the current pregnancy or postpartum
   6. Known severe hypertension (SBP >200mm/hg and/or DBP >120mm/hg) during the current pregnancy or postpartum
6. <18 years of age
7. Unable or refused consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | 6 months
  Mean recruitment rate per center per month

SECONDARY OUTCOMES:
Consent Rate | 6 months
  Proportion of eligible subjects who provide consent
Withdrawals/Loss to Follow-up | 9 months
  Proportion of withdrawals/loss to follow-up among participants
Study Drug Compliance | 6 months
  Level of compliance with study drug through participant recall and medication diary
Time Required to Obtain Site Institutional Approvals | 24 months
  Proportion of sites requiring >18 months to obtain all required approvals/contracts from time of delivery of all study documents.
VTE Event Rate | 6 months
  A more precise estimate of the VTE event rate
Bleeding Event Rate | 6 months
  A more precise estimate of the major and clinically relevant non-major bleeding event rate

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Skeith, MD, Principal Investigator — University of Calgary; Marc Rodger, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (7):
- Canada (4):
  - Foothills Medical Centre, Calgary, Alberta
  - British Columbia Women's Hospital & Health Centre, Vancouver, British Columbia
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
- Centre Hospitalier Universitaire de Saint-Etienne, Saint-Étienne-de-Montluc, Pays de la Loire Region, France
- Rotunda Hospital, Dublin, Ireland
- The Amsterdam Medical Centre, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Skeith L, Malinowski AK, El-Chaar D, Chan WS, Donnelly J, Chauleur C, Ganzevoort W, Wood S, Dubois S, McCarthy C, Buchmuller A, Wiegers H, Gibson PS, Ni Ainle F, Middeldorp S, Duffett L, Bates SM, Garven A, Baxter J, Lethebe BC, Rodger MA; Pilot PARTUM Group. Low-dose aspirin versus placebo in postpartum venous thromboembolism: a multi-national, pilot, randomised, placebo-controlled trial. Lancet Haematol. 2025 Feb;12(2):e109-e119. doi: 10.1016/S2352-3026(24)00338-7. Epub 2025 Jan 16. PMID 39827892
- [Derived] Blondon M, Claver M, Celetta E, Righini M, de Tejada BM. Preventing Postpartum Venous Thromboembolism With Low-Molecular-Weight Heparin: The PP-HEP Pilot Randomised Controlled Trial. BJOG. 2025 Jan;132(1):35-43. doi: 10.1111/1471-0528.17943. Epub 2024 Sep 5. PMID 39238110
- [Derived] Middleton P, Shepherd E, Gomersall JC. Venous thromboembolism prophylaxis for women at risk during pregnancy and the early postnatal period. Cochrane Database Syst Rev. 2021 Mar 29;3(3):CD001689. doi: 10.1002/14651858.CD001689.pub4. PMID 33779986